CLINICAL TRIAL: NCT05300334
Title: Prospective Observational Study Evaluating the Prevalence of Adenosine Deaminase (ADA) Enzyme Deficiency Disease in Lymphopenic Patients in Immunology Clinics
Brief Title: Investigation of ADA Enzyme Deficiency
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: TRPHARM (Industry)
Responsible Party: Sponsor
Other Study IDs: TR-ADA-002
Record Dates: First submitted 2022-03-18; First posted 2022-03-29 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Adenosine Deaminase Deficiency
Keywords: lymphopenia, adenosine deaminase, guithre paper
MeSH Terms: conditions — Severe combined immunodeficiency due to adenosine deaminase deficiency; Lymphopenia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: adenosine deaminase test — adenosine deaminase deficiency test

SUMMARY:
This observational study was designed as a prospective epidemiological screening study. Patients who applied to the centers participating in the study and were found to be lymphopenic in at least one examination will be included in the study. Up-to-date data will be collected from patients who have agreed to participate in the study, and a blood sample will be taken from patients on Guthrie paper. The blood taken will be sent to the Duzen Laboratories center located in Ankara and will be subjected to ADA metabolites analysis. For patients with a high metabolic test, the responsible investigator will advise on clarifying the diagnosis with a genetic test other than the study. In case of formation of new information for each patient, consultation will be provided by the responsible researcher. Thus, the prevalence of ADA enzyme deficiency disease in patients with lymphopenia will be evaluated. In addition, with this study, it will be scientifically demonstrated whether lymphopenia is a parameter that facilitates early diagnosis of ADA patients.

DETAILED DESCRIPTION:
Primary immune deficiencies present with signs and symptoms concerning the various disciplines of medicine when compared to other communities in our country on a more frequent basis and are determined severe combined immune deficiencies; T, B and NK cell development occasionally and/or errors caused by inherited genes that play a role in function, the immune system is a group of diseases of heterogeneous dysfunction that creates serious. The incidence is estimated at 1/100,000 live births in the United States. Although the exact incidence of inbreeding is not known in our country, where inbreeding is common, it is expected that those who show autosomal recessive transition will be more common, especially. Each step that is active in the emergence of an immune response creates the potential for a primary immunodeficiency disease. Due to the development of molecular and cellular techniques, the possibility of prenatal diagnosis has arisen with the detection of localization and mutations of the defective gene in various immunodeficiencies. The recognition of these disorders by clinicians is important for reducing long-term complications due to recurrent infections and preventing mortality with appropriate treatment. The frequency of SCID is not known in our country. Unlike in Europe and America, SCID types, which are autosomal recessive in our country, are considered to be the most common form due to high rates of inbreeding. The figure obtained by comparing the number of live babies born in a year in Konya with the number of SCID cases diagnosed in the Pediatric Immunology clinic of the Meram Faculty of Medicine of Selcuk University, the only primary immunodeficiency diagnostic center in the region, in the same year, is 1/10,000. This preliminary study shows that in our country this disease is much more common than in Europe and America. Based on the fact that about 1,400,000 babies are born per year in our country it should be expected that 140 new cases of SCID should be encountered every year. The number of cases diagnosed in our country is much lower than this figure. To date, more than 20 genetic defects have been identified that cause SCID. All known genetic defects disrupt the development of cells of the immune system, causing combined immunodeficiency. One of them, the ADA defect, is also a metabolic disease, due to which there is a lack of enzymes. ADA catalyzes the deamination of purine nucleosides adenosine (Ado) and 2'-deoxyadenosine (dAdo), which are produced during the degradation and transformation of RNA and DNA. ADA is a cleansing enzyme: it detoxifies purines. In ADA deficiency, 2'-deoxyadenosine (dAdo) is phosphorylated and converted into deoxyadenosine triphosphate (dATP). Accumulation of DATP disrupts DNA repair and replication. A high percentage of dATP accumulates in ADA deficiency, especially in erythrocytes and lymphocytes. Increased levels of adenosine break down the wall of the lymphocyte. It inhibits the development of lymphocytes in the thymus. A kind of lymphocyte intoxication occurs. It leads to a severe form of lymphopenia. Approximately 10-20% of SCID are diagnosed as ADA enzyme deficiency. It shows an autosomal recessive transition. Your gene is 20. it is localized on the long arm of the chromosome.

Clinically, there are early and late onset types. Classic-early onset ADA deficiency: Although normal at birth, patients present with infections seen from the first months of life, resulting in death if left untreated. In addition to the AKI table, neuro-developmental disorders, sensorineural hearing loss and/or skeletal abnormalities have also been reported in these patients. Although hematopoietic stem cell transplantation, enzyme replacement therapy and gene therapy are treatment approaches that provide cure, early diagnosis determines the prognosis. Late onset ADA deficiency: Patients may present with recurrent infections, autoimmunity, human papillomavirus (HPV) infections at an older age, even in adulthood. Lymphopenia is an invariable finding. High IgE and eosinophilia may be observed. In these cases, residual enzyme activity due to the type of mutation causes a late onset. This phenotype accounts for 10-15% of all cases of ADA deficiency. Diagnosis: ADA enzyme deficiency is included in severe combined immunodeficiencies and is observed with lymphopenia and infections. The diagnosis is made by measuring the activity of the enzyme ADA in erythrocytes or lymphocytes in patients with suspected clinical and laboratory features (such as lymphopenia). By mutation analysis, a gene defect is shown. However, T-cell receptor excision circles (TREC) test is used for early diagnosis. However, since the TREC test is found to be normal at birth in late-onset patients, screening that leads patients to an early diagnosis can only be achieved by measuring ADA metabolites. Although studies are continuing for SCID, which has not yet been included in the screening program in our country, the tandem mass spectrometer, which can be used to diagnose ADA deficiency, is used in newborn screening programs for metabolic diseases. Studies of newborn screening with a tandem mass spectrometer for ADA and PNP deficiencies, which is also a metabolic disease, began after 2010, and it has been shown that this method is a low-cost and reliable method. Early and late onset ADA deficiency cases can be detected with sensitivity and specificity reaching 100% with this method. Importance of early diagnosis: In Early Onset ADA deficiency, patients usually consult a doctor with signs of infections. The fact that infections are already common in the dairy childhood age group makes diagnosis difficult. If there is no similar case in the family that has been diagnosed before, or if this is not paid attention to in the history, the diagnosis of the cases is delayed. In late-onset ADA deficiency, the diagnosis is much more difficult. Low awareness of the disease and its symptoms usually results in these cases not being able to get a diagnosis, not being able to get effective treatment, and organ damage. For this reason, early diagnosis is very important in terms of quality of life as well as vital importance.

Grounds:

Data on the frequency of ADA enzyme deficiency in primary immunodeficiencies are insufficient. Because of the inability of these patients to get a diagnosis, their treatment is also inadequate. For the first time in our country, this study aims to determine the early diagnosis and obtain preliminary data on the prevalence of ADA disease by looking at ADA metabolites in the target patient group with lymphopenia and obtaining preliminary data on the prevalence of ADA disease.

ELIGIBILITY:
Inclusion Criteria:

1. Signing of the written informed consent form by the patient and/or his legal representative,
2. The presence of lymphopenia as a result of at least one hemogram of the patient,

   * The number of lymphocytes should be below 3000/mm3 for the first 0-12 months
   * The number of lymphocytes dec below 1500/mm3 for the first 13 months- ≤ 40 years
3. The patient should be 0- ≤ 40 years of age

Exclusion Criteria:

1. The patient was diagnosed with ADA enzyme deficiency before being included in the study,
2. The patient has participated in an interventional clinical trial within the last 30 days,
3. Failure of the patient himself and/or his legal representative to give their consent to participate in the study,
4. According to the researcher's opinion, the patient will not be able to properly fulfill the study requirements,
5. Pregnancy and/or lactation period
6. The fact that the volunteer participating in the study received an erythrocyte suspension or a complete blood transfusion within the last 3 months.

Max Age: 40 Years | Sex: All
Age Groups: Child, Adult
Study Population: 1. The presence of lymphopenia as a result of at least one hemogram of the patient,
     * The number of lymphocytes should be below 3000/mm3 for the first 0-12 months
     * The number of lymphocytes dec below 1500/mm3 for the first 13 months- ≤ 40 years
  2. The patient should be 0- ≤ 40 years of age
Sampling Method: Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2019-10-10 (Actual); Primary Completion 2020-11-05 (Actual); Study Completion 2022-10-10 (Estimated)

PRIMARY OUTCOMES:
The ratio of patients with a high ADA metabolite test to patients with lymphopenia | 2 years
  The proportion of patients with lymphopenia who have an ADA metabolite test above the threshold and are suspected of having an ADA enzyme deficiency

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Üniversitesi Tıp Fakültesi, Ankara, Mamak, Turkey (Türkiye)